CLINICAL TRIAL: NCT01896648
Title: Sexual Dysfunction in Type 2 Diabetic Women: Study on Prevalence and on Risk
Brief Title: Sexual Dysfunction in Type 2 Diabetic Women
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Professor, University of Pavia
Other Study IDs: 20120021266
Record Dates: First submitted 2013-06-25; First posted 2013-07-11 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Sexual Dysfunction; Neuropathy
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — The following parameters will be assessed:
  Blood: ematology, glycated hemoglobin, fasting plasma glucose, fasting plasma insulin, total cholesterol, HDL cholesterol, triglycerides, LDL cholesterol, creatinine, urea, transaminases, electrolytes, homocysteine, high sensitivity C-reactive protein (hs-CRP), metalloproteinase-2 (MMP-2), metalloproteinase-9 (MMP-9), soluble adhesion molecules (sICAM-1, sVCAM-1), sE-selectin, lipoprotein (a) [Lp (a)], Plasminogen Activator Inhibitor-1 (PAI-1).
  Urine: complete urinalysis, 24-hour microalbuminuria
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 2 diabetic women

SUMMARY:
Type 2 diabetes mellitus is becoming an increasingly problem for public health and it is related with various complications such as sexual problems. The prevalence of erectile dysfunction has been widely studied in men as a complication of diabetes; the prevalence of sexual dysfunction in women, instead, has not been well investigated. The aim of this study is to evaluate the prevalence of sexual dysfunction in type 2 diabetic women using international validated questionnaires.

DETAILED DESCRIPTION:
In an estimated temporal space of about 3 years, 306 women will be recruited consecutively.

After collection of written informed consent, the following data will be collected:

* History: type of diabetes, comorbidities, current medication, duration of diabetes and complications, voluptuary habits such as tobacco smoke (both number of packets/year and n° packets/day), alcohol consumption, coffee consumption, physical activity.
* Physical exam, general anthropometric parameters such as weight, height, circumference, body mass index, waist-hip ratio, and blood pressure.
* Assessment of glycemic variability (fasting plasma glucose and post-prandial glucose)
* Each patient will be self-administered Female Sexual Function Index (FSFI) and Female Sexual Distress Scale (FSDS) questionnaires to assess the prevalence of sexual dysfunction and Self-Rating Anxiety Scale (SAS) and Self-Rating Depression Scale (SDS) of Zung for an accurate assessment of the state of anxiety and depression.
* We will collect blood and urine samples to assess: ematology, glycated hemoglobin, fasting plasma glucose, fasting plasma insulin, total cholesterol, HDL cholesterol, triglycerides, LDL cholesterol, creatinine, urea, transaminases, electrolytes, complete urinalysis, 24-hour microalbuminuria, homocysteine, high sensitivity C-reactive protein (hs-CRP), metalloproteinase-2 (MMP-2), metalloproteinase-9 (MMP-9), soluble adhesion molecules (sICAM-1, sVCAM-1), sE-selectin, lipoprotein (a) [Lp (a)], Plasminogen Activator Inhibitor-1 (PAI-1).
* We will also conduct a clinical and instrumental exam of the foot using Neuropad, recently validated as a screening tool for diabetic neuropathy. Patients will also undergo autonomic tests (deep breathing, lying to standing, Valsalva maneuver, and orthostatic hypotension).

We will also evaluate the presence of neuropathy through the administration of the Michigan Neuropathy Screening Instrument (MNSI) and the Neuropathy Disability Score (NDS).

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus

Exclusion Criteria:

* previous surgery for hysterectomy or ovariectomy
* hormone replacement

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic women
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2013-06-24 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) | 12 months
  Female Sexual Function Index (FSFI) is a 19-item questionnaire, developed as a brief, multidimensional self-report instrument for assessing the key dimensions of sexual function in women.

SECONDARY OUTCOMES:
Prevalence of sexual dysfunction risk factors | 36 months
  We will consider the following risk factors:
  Smoking status; Consume of alcohol; Obesity; Hepatic steatosis; Hypertension; Dyslipidemia; Chronic ischemic disease; Hyperuricemia; Chronic kidney disease; Retinopathy; Neuropathy; Vasculopathy.
  Correlations between sexual dysfunction and single risk factors will be analyzed using the Pearson correlation coefficient r.

OTHER OUTCOMES:
Correlation between sexual dysfunction and diabetic neuropathy | 36 months
  The presence of diabetic neuropathy will be assessed using dysautonomic tests (deep breathing, lying to standing, Valsalva maneuver e orthostatic hypotension).
  The prevalence of symmetric distal neuropathy will be assessed using:
  1. the Neuropad test, developed as a simple visual indicator test to evaluate diabetic neuropathy
  2. the Michigan Neuropathy Screening Instrument (MNSI)
  3. the Neuropathy Disability Score (NDS) The correlation will be analyzed using the Pearson correlation coefficient r

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Derosa, MD, PhD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia
Locations (1):
- IRCCS Policlinico S. Matteo Foundation, Pavia, Italy